CLINICAL TRIAL: NCT06810362
Title: Walking Our Way to a Healthier Brain: a Randomized Controlled Trial to Evaluate the Effects of Aerobic Exercise, Cognitive Remediation and Combined Intervention in Schizophrenia
Brief Title: Effects of Aerobic Exercise, Cognitive Remediation and Combined Intervention in Schizophrenia
Acronym: C-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marta Bosia, Prof.ssa, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2016-02361538
Record Dates: First submitted 2025-01-09; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia; Psychosis
Keywords: cognition; pshysical activity; metabolic syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Metabolic Syndrome | interventions — Cognitive Remediation; Exercise

STUDY DESIGN:
Intervention Model Description: All patients will be randomized in a 1:1:1 ratio to three parallel treatment arms: experimental intervention (CR + AE) and two active comparison arms (CR and AE)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive Remediation (CR) (Active Comparator): CR consists of three 1-hour sessions per week of domain-specific computerized exercises, over a 12-week period, for a total of 36 hours
  Interventions: Behavioral: Cognitive Remediation (CR); Other: Cognitve Remediation + Aerobic Exercise
- Aerobic Exercise (AE) (Active Comparator): AE consists of 45 minutes of cycling twice a week, with 15 minutes of warm up pre and post session
  Interventions: Behavioral: Aerobic Exercise; Other: Cognitve Remediation + Aerobic Exercise
- Cognitive Remediation and Aerobic Exercise (Experimental): this intervention is composed by both cognitive remediation and aerobic exercise
  Interventions: Behavioral: Cognitive Remediation (CR); Behavioral: Aerobic Exercise; Other: Cognitve Remediation + Aerobic Exercise

INTERVENTIONS:
Behavioral: Cognitive Remediation (CR) — The CR consists of three 1-hour sessions per week of domain-specific computerized exercises, for a period of 12 weeks, totaling 36 hours
  Arms: Cognitive Remediation (CR); Cognitive Remediation and Aerobic Exercise
Behavioral: Aerobic Exercise — Aerobic exercise consists in two session per week of cycling. Each session lasts for 45 min, with 15 min of warm up pre and post session
  Arms: Aerobic Exercise (AE); Cognitive Remediation and Aerobic Exercise
Other: Cognitve Remediation + Aerobic Exercise — Patients performed both CR exercises and cycling

SUMMARY:
Tracking down the efficacy of a combined intervention of cognitive remediation (CR) and phisycal activity (aerobic exercise, AE) in patients diagnosed with schizophrenia

DETAILED DESCRIPTION:
The investigators will address the following objectives:

* Primary objective: o assess, through a randomized controlled trial (RCT), the efficacy and feasibility of a combined intervention (CR + AE) in patients with schizophrenia. The primary outcome measure will be cognitive performance, while secondary outcomes will include scales for the assessment of psychopathology, daily functioning, and quality of life.
* Secondary objectives: to evaluate changes in bio-physical and laboratory metabolic parameters, as well as in neurotrophic and neuroinflammatory factors. Furthermore, multimodal magnetic resonance imaging (MRI) parameters will be evaluated after the interventions, and their relationship with observed cognitive improvements will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Schizophrenia
2. Age 18-65 years
3. Psychopathological stability
4. Ability to provide informed consent

Exclusion Criteria:

1. Comorbidity with intellectual disability and neurological disorders.
2. Ongoing treatment with CR or AE.
3. Specific contraindications for AE.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 7 months
  Cognition is assessed through the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB): a neuropsychological battery developed for the assessment of the main cognitive domains impaired in schizophrenia. Range T-values: 20-80. Higher values mean a better score

SECONDARY OUTCOMES:
Psychopathology assessment | 7 months
  Psychopathology is assessed trough the scale Positive and Negative Syndrome Scale (PANSS). Values range 1-7, higher scores mean worse functioning
Quality of Life assessment | 7 months
  Quality of life is assessed through the scale Quality of Life Scale (QLS). Values range 0-6. Higher values mean better functioning
Daily functioning assessment | 7 months
  daily functioning is assessed through the task UCSD Performance-based skill assessment (UPSA-B). Values range 0-1. 1 means better functioning
Body Mass Index (BMI) | 7 months
  Physical fitness is assessed through the evaluation of BMI (kg/m^2)
Diffusion Tensor Imaging (DTI) | 4 months
  DTI was performed to assess the integrity of brain white matter and to estimate the axonal organization of the brain. Its unit of measure is µm²/ms
Waist circumference | 7 months
  Waist circumference (cm) is assessed for the evaluation of physical fitness
Blood pressure | 7 months
  Systolic and diastolic blood pressure (mm Hg) are assessed for the evaluation of metabolic syndrome and physical fitness
Metabolic indices | 7 months
  Tryglicerides, HDL cholesterol and fasting plasma glucose are assessed through blood sampling. All of them are measured in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Marta Bosia, MD, PhD, Principal Investigator — Vita-Salute San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinrichs DW, Hanlon TE, Carpenter WT Jr. The Quality of Life Scale: an instrument for rating the schizophrenic deficit syndrome. Schizophr Bull. 1984;10(3):388-98. doi: 10.1093/schbul/10.3.388. PMID 6474101
- [Background] Mausbach BT, Harvey PD, Goldman SR, Jeste DV, Patterson TL. Development of a brief scale of everyday functioning in persons with serious mental illness. Schizophr Bull. 2007 Nov;33(6):1364-72. doi: 10.1093/schbul/sbm014. Epub 2007 Mar 6. PMID 17341468
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Cavallaro R, Anselmetti S, Poletti S, Bechi M, Ermoli E, Cocchi F, Stratta P, Vita A, Rossi A, Smeraldi E. Computer-aided neurocognitive remediation as an enhancing strategy for schizophrenia rehabilitation. Psychiatry Res. 2009 Oct 30;169(3):191-6. doi: 10.1016/j.psychres.2008.06.027. Epub 2009 Sep 9. PMID 19740550
- [Background] Cassilhas RC, Tufik S, de Mello MT. Physical exercise, neuroplasticity, spatial learning and memory. Cell Mol Life Sci. 2016 Mar;73(5):975-83. doi: 10.1007/s00018-015-2102-0. Epub 2015 Dec 8. PMID 26646070
- [Background] Firth J, Cotter J, Elliott R, French P, Yung AR. A systematic review and meta-analysis of exercise interventions in schizophrenia patients. Psychol Med. 2015 May;45(7):1343-61. doi: 10.1017/S0033291714003110. Epub 2015 Feb 4. PMID 25650668
- [Background] Bryce S, Sloan E, Lee S, Ponsford J, Rossell S. Cognitive remediation in schizophrenia: A methodological appraisal of systematic reviews and meta-analyses. J Psychiatr Res. 2016 Apr;75:91-106. doi: 10.1016/j.jpsychires.2016.01.004. Epub 2016 Jan 5. PMID 26828372
- [Background] Laursen TM, Munk-Olsen T, Vestergaard M. Life expectancy and cardiovascular mortality in persons with schizophrenia. Curr Opin Psychiatry. 2012 Mar;25(2):83-8. doi: 10.1097/YCO.0b013e32835035ca. PMID 22249081
- [Background] Bowie CR, Reichenberg A, Patterson TL, Heaton RK, Harvey PD. Determinants of real-world functional performance in schizophrenia subjects: correlations with cognition, functional capacity, and symptoms. Am J Psychiatry. 2006 Mar;163(3):418-25. doi: 10.1176/appi.ajp.163.3.418. PMID 16513862
- [Background] Malchow B, Keeser D, Keller K, Hasan A, Rauchmann BS, Kimura H, Schneider-Axmann T, Dechent P, Gruber O, Ertl-Wagner B, Honer WG, Hillmer-Vogel U, Schmitt A, Wobrock T, Niklas A, Falkai P. Effects of endurance training on brain structures in chronic schizophrenia patients and healthy controls. Schizophr Res. 2016 Jun;173(3):182-191. doi: 10.1016/j.schres.2015.01.005. Epub 2015 Jan 23. PMID 25623601
- [Background] Penades R, Pujol N, Catalan R, Massana G, Rametti G, Garcia-Rizo C, Bargallo N, Gasto C, Bernardo M, Junque C. Brain effects of cognitive remediation therapy in schizophrenia: a structural and functional neuroimaging study. Biol Psychiatry. 2013 May 15;73(10):1015-23. doi: 10.1016/j.biopsych.2013.01.017. Epub 2013 Feb 26. PMID 23452665